CLINICAL TRIAL: NCT03429452
Title: Population-based Study to Identify Structural Heart Disease Abnormalities in a Spanish Community: Salamanca. The SALMANTICOR Study
Brief Title: The SALMANTICOR Study
Acronym: SALMANTICOR
Status: Completed | Type: Observational
Sponsor: AORTICA Group (Other)
Collaborators: University of Salamanca (Other)
Responsible Party: Principal Investigator, Pedro L Sanchez, Head of Cardiology, PhD, MD, Salamanca University Hospital
Other Study IDs: PI14/00695
Record Dates: First submitted 2018-01-10; First posted 2018-02-12 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Structural Heart Abnormality
Keywords: structural heart abnormality; spatial method; echocardiography; electrocardiogram; mediterranean diet; exercise; social status; rural
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Biomarkers and DNA samples will be stored in a biobank
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SALMANTICOR study will obtain data on the prevalence and incidence of structural heart disease in a population setting. A cross-section survey of randomly selected residents of Salamanca (Spain) will be performed. A total of approximately 2400 individuals, stratifies by place of residence (rural and urban) and by age and sex will be studied. The variables to analyzed will be obtained from the clinical history, different surveys including social status, Mediterranean diet, functional capacity, electrocardiogram, echocardiogram and biochemical and genetic analysis. Surviving participants are expected to return for a 5 and 10-year follow-up visit.

DETAILED DESCRIPTION:
The objectives of this study are: to obtain data on the prevalence and incidence of structural heart disease in a population setting; to show the spatial distribution different patterns of structural heart disease through the spectrum of age and sex and between urban and rural; and to generate new hypotheses which might serve to healthcare research and to political commitment to obtain resources and support effective public health program implementation.

The SALMANTICOR study is a cross-sectional descriptive population-based study of the prevalence of structural heart disease and their risk factors that will enroll a total of 2400 individuals, stratifies by place of residence (rural and urban), by age and by sex, in a Spanish community: Salamanca. Cohort participants will undergo a basal examination visit between 2015 and 2018. Surviving participants are expected to return for a 5 and 10-year follow-up visit. Institutional review committee approval was obtained and all participants will provide informed consent. The SALMANTICOR study is designed to provide echocardiographic parameters characterizing cardiac structure and function in all individuals. Medical history, surveys completion, and examinations will be obtained at the subject´s primary care referral center and will be analyzed and interpreted centrally at University Hospital of Salamanca. A complete medical history, physical examination and the surveys completion checkout will be performed by a cardiologist in a separate office to where examinations and blood sample extraction will be performed. Echocardiographic measures will be initially performed. Participant blood pressure and VASERA measures will be taken within 30 minutes of starting the echocardiographic exam and after the subject will be resting for 10 minutes. ECG will be performed after VASERA to finalize with the blood sample extraction. A magnetic resonance substudy and and a details analyses in diabetic individuals will also performed. SALMANTICOR participants will undergo surveillance for cardiovascular events, including heart failure, incident coronary heart disease, and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Any individual willing to participate

Exclusion Criteria:

* Death people not identified in the community records
* Not able to attend the visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2400 individuals, stratifies by place of residence (rural and urban), by age and by sex, in a Spanish community: Salamanca
Sampling Method: Probability Sample
Enrollment: 2057 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
prevalence of structural heart disease in a population setting | through study completion, an average of 3 years
  Structural heart disease refers to any of the following heat abnormalities including congenital heart disease, cardiomyoptathies, valvular heart disease, pericardial diseases and rhythm or conduction disorders
incidence of structural heart disease in a population setting | 5 years follow-up
  Structural heart disease refers to any of the following heat abnormalities including congenital heart disease, cardiomyoptathies, valvular heart disease, pericardial diseases and rhythm or conduction disorders

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Melero-Alegria JI, Cascon M, Romero A, Vara PP, Barreiro-Perez M, Vicente-Palacios V, Perez-Escanilla F, Hernandez-Hernandez J, Garde B, Cascon S, Martin-Garcia A, Diaz-Pelaez E, de Dios JM, Uribarri A, Jimenez-Candil J, Cruz-Gonzalez I, Blazquez B, Hernandez JM, Sanchez-Pablo C, Santolino I, Ledesma MC, Muriel P, Dorado-Diaz PI, Sanchez PL. SALMANTICOR study. Rationale and design of a population-based study to identify structural heart disease abnormalities: a spatial and machine learning analysis. BMJ Open. 2019 Feb 13;9(2):e024605. doi: 10.1136/bmjopen-2018-024605. PMID 30765403